CLINICAL TRIAL: NCT03700372
Title: IMPACT: A Safety and Feasibility Study of the IOWA Approach Cardiac Ablation System
Acronym: IMPACT
Status: Completed | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0172
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-08

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients with paroxysmal atrial fibrillation undergoing cardiac surgery and meeting all protocol inclusion/exclusion criteria will be treated with the IOWA Approach Cardiac Ablation System.
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (1):
- IOWA Approach Cardiac Ablation (Experimental): Subjects who are treated with the IOWA Approach Cardiac Ablation System for paroxysmal atrial fibrillation.
  Interventions: Device: IOWA Approach Cardiac Ablation System

INTERVENTIONS:
Device: IOWA Approach Cardiac Ablation System — Epicardial ablation using the IOWA Approach Cardiac Ablation System

SUMMARY:
IMPACT is a prospective, single-arm, multi-center, safety and feasibility study evaluating the IOWA Approach Cardiac Ablation System (FARAPULSE, Inc.) for the treatment of paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
Patients with paroxysmal atrial fibrillation scheduled to undergo cardiac surgery will be screened for enrollment per protocol inclusion and exclusion criteria. Enrolled patients will then undergo ablation using the IOWA Approach Cardiac Ablation System (FARAPULSE, Inc.), followed by concomitant cardiac surgery. Subjects will be followed at 7 days, 30 days, 3 months, 6 months and 12 months with a blanking period for recurrent atrial fibrillation or atrial tachycardia of 3 months following the index ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥ 18 and ≤ 70 years of age on the day of enrollment.
2. Diagnosis of paroxysmal atrial fibrillation defined as symptomatic paroxysmal AF with at least two episodes of paroxysmal AF observed within the 12 months preceding inclusion.
3. Patients are resistant to anti-arrhythmic treatments.
4. Anteroposterior Left atrial diameter ≤ 5.5 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT) within 3 months prior to the procedure.
5. Subject has no contraindications to intraoperative transesophageal echocardiography;
6. Subject is scheduled to undergo elective on-pump cardiac surgical procedure(s) to be performed including open-heart surgery for one or more of the following:

   * Mitral valve repair or replacement,
   * Aortic valve repair or replacement
   * Tricuspid valve repair or replacement, or
   * Coronary artery bypass procedures
7. Left ventricular ejection fraction ≥40% as documented by TTE within 12 months prior to the procedure.
8. Received a standard cardiac work up and is an appropriate candidate for an investigational procedure as determined by trial investigators.
9. Subject is willing and capable of providing Informed Consent to undergo study procedures and participate in all examinations and follow-ups associated with this clinical trial.

Exclusion Criteria:

1. Abnormal cardiac and/or epicardial anatomy (such as adhesion, anomalous coronaries, thickened epicardium, etc.) or pericardial reflections on TTE, MRI or CT.
2. Prior left-sided cardiac ablation.
3. Prior history of open chest surgery and/or any procedure where the pericardial space was entered or instrumented (pericardiocentesis, catheter mapping and /or ablation).
4. Patient has a prosthetic heart valve.
5. Patient has a left atrial appendage device
6. Prior history of pericarditis or pericarditis within 3 months based on the TTE examination.
7. Subject is a woman of child bearing age
8. Prior history of rheumatic fever.
9. Prior history of medical procedure involving instrumentation of the left atrium (previous ablation, Atrial septal defect) ASD closure, left atrial appendage occlusion)
10. History of severe chronic gastrointenstinal problems involving the esophagus, stomach and/or untreated acid reflux
11. History of abnormal bleeding and/or clotting disorder.
12. Active malignancy or history of treated cancer within 24 months of enrollment.
13. Clinically significant infection or sepsis.
14. History of stroke or TIA within prior 6 months
15. New York heart Association (NYHA) class IIIb or IV congestive heart failure and/or any heart failure hospitalization within 3 months prior to enrollment.
16. Body mass index > 35.
17. Estimate glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 or has ever received dialysis.
18. History of untreated and serious hypotension, bradycardia or chronotropic incompetence.
19. Any of the following within 3 months of enrollment:

    * Major surgery except for the index procedure
    * Myocardial infarction
    * Unstable angina
    * Percutaneous coronary intervention (e.g., CABG or PTCA)
    * Sudden cardiac death event
    * Left atrial thrombus that has not resolved as shown by TEE (transesophageal echo) or CT
    * Implant of pacemaker, ICD (implantable cardioverter defribillator) or CRT (cardiac resynchronization therapy).
20. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
21. History of pulmonary hypertension with Pulmonary systolic artery pressure >50 mm Hg, severe Chronic Obstructive Pulmonary Disease or restrictive lung disease.
22. Patients with any other significant uncontrolled or unstable medical condition (such as uncontrolled brady-arrhythmias, ventricular arrhythmias, hyperthyroidism or significant coagulation disorder).
23. Life expectancy less than one year.
24. Clinically significant psychological condition that in the physician's opinion would prohibit the subject's ability to meet the protocol requirements.
25. Enrolled in another cardiac clinical trial that would interfere with this trial.
26. Life expectancy less than one year.
27. Clinically significant psychological condition that in the physician's opinion would prohibit the subject's ability to meet the protocol requirements.
28. Enrolled in another cardiac clinical trial that would interfere with this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2021-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Single Arm Study
Period: Overall Study
Arm/Group | IOWA Approach Cardiac Ablation
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IOWA Approach Cardiac Ablation
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: Years] | 69 [63 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 4
  France | 3

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety: A Composite Safety Endpoint Consisting of the Subjects That Experience One or More Serious Adverse Events (SAEs) Related to the Investigational Procedure and/or Device Within 30 Days of the Ablation Procedure or Hospital Discharge.
Description: A composite safety endpoint consisting of the proportion of subjects that experience one or more of the following serious adverse events (SAEs) related to the investigational procedure and/or device within 30 days of the PEF (pulsed electric field) ablation procedure or hospital discharge, whichever is later, except as noted below:
  * Cardiac death
  * Stroke and/or transient ischemic attack (TIA)
  * Myocardial infarction (MI)
  * Excessive bleeding
  * Atrio-esophageal fistula
  * Persistent post-surgical phrenic nerve paralysis at 12 months
  * Severe pulmonary vein stenosis (>70%)
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | IOWA Approach Cardiac Ablation
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Feasbility: Electrical Isolation of Posterior Left Atrium and Pulmonary Veins.
Description: Proportion of subjects that achieve procedural success. Procedural success is defined as the creation of an electrically isolating "box" lesion encompassing the pulmonary veins and posterior left atrium using the study device.
Time Frame: 1 Day (Acute)
Measure: Count of Participants; unit: Participants
Arm/Group | IOWA Approach Cardiac Ablation
Number analyzed (Participants) | 7
Participants | 6

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | IOWA Approach Cardiac Ablation
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IOWA Approach Cardiac Ablation (N=7)
Hematoma (Vascular disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Malaise (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IOWA Approach Cardiac Ablation (N=7)
Paroxysmal Fibrillation (Cardiac disorders) | 2 (2)
Vertigo (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Pain and redness in the sternotomy area (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Swelling of lower limbs (Vascular disorders) | 3 (3)
Dyspnea (Nervous system disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Numbness of lower limb (Vascular disorders) | 1 (1)
Tumor in pulmonary region (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematuria post-surgery (Vascular disorders) | 1 (1)
Atrial fibrillation recurrence (Cardiac disorders) | 1 (1)
Visual disorder (Eye disorders) | 2 (2)
insomnia (General disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bloody Spittle (General disorders) | 1 (1)
Vagal discomfort without loss of consciousness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: CS0172-001 (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT03700372/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: CS0172-002 (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT03700372/Prot_SAP_003.pdf